CLINICAL TRIAL: NCT05552105
Title: The Oxylipin Response as a New PrEdictive Biomarker of Patient Responsiveness to Biotherapy in Rheumatoid Arthritis.
Brief Title: The Oxylipin Response as a New PrEdictive Biomarker of Patient Responsiveness to Biotherapy in Rheumatoid Arthritis (OPERA)
Acronym: OPERA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other); University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: RBHP 2022 TOURNADRE
Record Dates: First submitted 2022-09-16; First posted 2022-09-23 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Anti TNF; Oxylipin; Cytokine; Polyunsatured fatty acid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort (Other)
  Interventions: Other: Blood test

INTERVENTIONS:
Other: Blood test — Before and after 6-months of anti TNF treatment, blood will be collected using the TruCulture system (2x 1ml in non-stimulated and LPS-stimulated TruCulture tubes) to measure Whole Blood Oxylipin Response, cytokine response, PUFA cell content and gene expression under homeostatic and stimulated conditions (i.e. LPS)

SUMMARY:
OPERA aims to better understand and predict the responsiveness of rheumatoid arthrits (RA) patients to biological disease modifying anti-rheumatic drugs (bDMARDs).

Our objectives will be (i) to determine, at baseline, the differences of oxylipin response between responders vs non-responders to Anti-Tumor necrosis factor (Anti TNF) and (ii) to investigate the relationships between the oxylipin response, the polyunsatured fatty acid (PUFA) content of immune cells and the cytokine response.

DETAILED DESCRIPTION:
30 RA patients starting an anti-TNF will be recruited.

Before and after 6-months of anti-TNF treatment, blood will be collected using the TruCulture system (2x 1ml in non-stimulated and Lipopolysaccharide (LPS)-stimulated TruCulture tubes) to measure Whole Blood Oxylipin Response (WBOR), cytokine response, PUFA cell content and gene expression under homeostatic and stimulated conditions (i.e. LPS).

At baseline and after 6 months of treatment, the rheumatologist will perform a clinical evaluation of their RA patients using Disease Activity Score using 28 joint-count (DAS28-CRP). Non-responders will be defined as RA patients failing to achieve good or moderate EULAR response after 6 month of anti-TNF treatment, discontinued the drug, initiated a new bDMARD, or increased dosage of oral corticosteroids greater than 10 mg/d at the second visit.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid patient according to ACR-EULAR (American college of rheumatology-European League Against Rheumatism) 2010 criteria,
* Active disease defined by a DAS28-CRP>3.2,
* Biological and targeted synthetic DMARDs naïve,
* Indication for treatment with anti-TNF
* Stable corticosteroid therapy ≤ 10 mg/day

Exclusion Criteria:

* Contra-indications to a biological DMARDS (current or recent cancer, active infection),
* Non-steroidal anti-inflammatory drugs (NSAIDs) treatment during the last 2 weeks before inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2025-01-28 (Actual); Study Completion 2025-01-28 (Actual)

PRIMARY OUTCOMES:
Quantification of total oxylipins | Baseline
  Quantitative profiling procedure for oxylipins

SECONDARY OUTCOMES:
Quantification of polyunsatured fatty acids in blood cells | Baseline
  Quantitative profiling procedure for polyunsatured fatty acids in blood cells (leukocytes, red blood cells and platelets)
Quantification of cytokines | Baseline
  Large panel of 21 cytokines characteristic of the inflammatory response and lymphocyte polarization. (IL-1β, IFN-α2, IFN-γ, TNF-α, MCP-1 (CCL2), IL-6, IL-8 (CXCL8), IL-10, IL-12p70, IL-17A, IL-18, IL-23, IL-33, IL-5, IL-13, IL-2, IL-9, IL-10, IL-17F, IL-4, IL-22)
EULAR Response | 6 month
  Non-responders will be defined as rheumatoid arthritis patients failing to achieve good or moderate EULAR response after 6 month of biological disease modifying anti rheumatic drug (bDMARD), discontinued the drug, initiated a new bDMARD, or increased dosage of oral corticosteroids greater than 10 mg/d at the second visit.
  EULAR response is determined by the decrease in Disease activity score (DAS) between Baseline and 6 months
Quantification of total oxylipins | 6 month
  Quantitative profiling procedure for oxylipins
Quantification of cytokines | 6 month
Quantification of polyunsatured fatty acids in blood cells | 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No